CLINICAL TRIAL: NCT07183800
Title: Does a 10-minute Trampoline Protocol Induce Urine Leakage or Changes in Pelvic Morphometry Among Females Who Report That They do Not Experience Symptoms of Urinary Incontinence?
Brief Title: Trampoline-Induced Changes in Pelvic Structure and Continence
Acronym: TRAM
Status: Recruiting | Type: Observational
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Linda McLean, Full Professor, University of Ottawa
Other Study IDs: H-05-25-11551
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Urinary Continence; Urinary Incontinence; Urinary Incontinence (UI); Urinary Incontinence , Stress
Keywords: stress urinary incontinence; pelvic floor; pelvic floor morphology; high impact exercise; urine leakage; urinary symptoms; levator plate; female athletes; bladder neck; posterior urethro-vesical angle; PUVA; jump; trampoline; high impact; high intensity; healthy female; incontinence; leakage; urinary leakage
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress | interventions — Water

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy young active females: 18-40yo active females with no self-reported urinary incontinence
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Participants will undergo a standardized 10-minute high-intensity trampoline jumping protocol designed to elicit mechanical loading on the pelvic floor. Prior to the jumping session, bladder volume will be assessed via transabdominal ultrasound. If a participant's bladder contains less than 100 mL of urine, they will be asked to drink water and wait until a target range of 100-200 mL is reached to ensure consistent pre-jump bladder filling across participants. This approach minimizes variability in bladder volume, which could influence pelvic floor measurements.

SUMMARY:
The goal of this clinical trial is to evaluate whether a short bout of high-intensity trampoline jumping induces urinary leakage or measurable changes in pelvic floor morphology in active females aged 18-40 who do not report symptoms of urinary incontinence. The main questions it aims to answer are:

Hypothesis 1: Does a single 10-minute trampoline protocol result in acute changes in pelvic floor structure, including bladder neck position, levator plate length, and/or posterior urethrovesical angle (PUVA)?

Hypothesis 2: Do participants report any urinary leakage during the jumping protocol, despite being asymptomatic at baseline?

Hypothesis 3: Do pelvic morphology changes recover within 30 minutes post-jumping, or do alterations persist?

Researchers will perform within-subject comparisons at multiple time points (pre-jump, immediately post-jump, and 30 minutes post-jump) using transperineal ultrasound imaging to assess structural changes.

Participants will:

* Attend one laboratory visit
* Complete baseline pelvic health questionnaires (ICIQ-UI Short Form and PFD Sentinel).
* Undergo 2D transperineal ultrasound imaging in the standing position at rest, immediately post-jumping, and 30 minutes post-jumping.
* Perform a 10-minute high-intensity jumping protocol on a mini-trampoline, while heart rate and perceived exertion are monitored.
* Verbally report any urine leakage during jumping using standardized descriptors.

DETAILED DESCRIPTION:
Urinary incontinence (UI) has traditionally been associated with postpartum or older women; however, growing evidence highlights its prevalence among young, physically active females - even in those without a history of pelvic floor dysfunction or childbirth. High-impact physical activities such as running, jumping, and trampolining have been shown to increase intra-abdominal pressure, placing acute mechanical stress on the pelvic floor and potentially contributing to urinary leakage. While the relationship between high-impact exercise and stress urinary incontinence (SUI) has been explored in terms of prevalence, less is known about the acute, real-time mechanical effects of impact loading on pelvic floor structures in asymptomatic individuals.

This study aims to investigate whether a 10-minute high-intensity trampoline protocol induces measurable changes in pelvic morphology - specifically in bladder neck position, levator plate length, and/or posterior urethrovesical angle (PUVA) - in physically active females aged 18-40 who do not report urinary incontinence symptoms. These anatomical parameters are indicators of pelvic floor support and dysfunction, and their change under load may signal early mechanical strain on the pelvic floor.

Participants will undergo a single study session involving a baseline transperineal ultrasound assessment, a 10-minute jumping bout, and follow-up ultrasound assessments immediately, and 30 minutes post-exercise. Urinary leakage is monitored during jumping via verbal self-report every 2 minutes, with descriptive classifications such as "drops," "squirt," or "gush." Jumping intensity is tracked using the Borg RPE scale and heart rate monitoring via Apple Watch, which has demonstrated acceptable validity for exercise heart rate tracking.

A repeated-measures design will be used to assess within-subject changes in pelvic morphology, with participants serving as their own control across time points. Data will be analyzed using repeated-measures ANOVA to determine statistically significant changes, with Cohen's d effect sizes calculated to assess magnitude of effect. Leakage data will be reported descriptively.

Ultimately, this study will generate foundational data on the immediate biomechanical response of the pelvic floor to high-impact activity. These findings may help identify early indicators of pelvic floor strain, even in women without symptomatic UI, and could inform future screening and prevention strategies for active female populations.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40
* Engage in regular physical activity or sport
* Do not experience frequent urinary leakage (no more than once per month during exercise, coughing, or sneezing)
* Can complete a 10-minute jumping protocol

Exclusion Criteria:

* Currently pregnant or have been pregnant in the past 6 months
* Have cardiac, pulmonary, metabolic, and/or neurological conditions
* Have a lower body injury that limits your ability to jump
* Have had a hysterectomy and/or incontinence surgery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited from the Ottawa region through local gyms, university facilities, and social media platforms. The study population includes recreationally active females aged 18-40 who engage in activities such as running or brisk walking and are willing to attend a single in-person session at the University of Ottawa's Motor Function Measurement Laboratory.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessing whether a short-duration trampoline protocol induces urinary leakage in active females. | Urinary leakage is assessed during the 10-minute jumping protocol on the single lab visit.
  Urinary leakage is assessed via self-report during a 10-minute high-intensity trampoline jumping protocol. Every 2 minutes, participants are verbally prompted to report whether they experienced leakage, and to classify it using standardized descriptors ("drops," "squirt," or "gush"). Leakage severity is indexed based on the timing of first report, frequency of episodes, and qualitative volume descriptors. Descriptive statistics will be used to report the proportion of participants who leak, frequency of leakage, and severity profiles.

SECONDARY OUTCOMES:
Assessing whether a short-duration trampoline protocol induces acute changes in bladder neck morphology in active females. | Bladder neck morphology outcomes are assessed across a single session spanning approximately 45-60 minutes (baseline through 30 minutes post-exercise).
  Bladder neck morphology is measured at three time points (pre-jumping, immediately post-jumping, and 30 minutes post) using 2D transperineal ultrasound imaging. Repeated-measures ANOVA will be used to determine significant changes in bladder neck morphology across time points. Cohen's d effect sizes will be calculated to assess the magnitude of observed changes.
Assessing whether a short-duration trampoline protocol induces acute changes in levator plate length in active females. | Levator plate length outcomes are assessed across a single session spanning approximately 45-60 minutes (baseline through 30 minutes post-exercise).
  Levator plate length is measured at three time points (pre-jumping, immediately post-jumping, and 30 minutes post) using 2D transperineal ultrasound imaging. Repeated-measures ANOVA will be used to determine significant changes in levator plate length across time points. Cohen's d effect sizes will be calculated to assess the magnitude of observed changes.
Assessing whether a short-duration trampoline protocol induces acute changes in the posterior urethrovesicle angle (PUVA) in active females. | Posterior urethrovesicle angle (PUVA) outcomes are assessed across a single session spanning approximately 45-60 minutes (baseline through 30 minutes post-exercise).
  The posterior urethrovesicle angle (PUVA) is measured at three time points (pre-jumping, immediately post-jumping, and 30 minutes post) using 2D transperineal ultrasound imaging. Repeated-measures ANOVA will be used to determine significant changes in the PUVA across time points. Cohen's d effect sizes will be calculated to assess the magnitude of observed changes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa - Lees Campus, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Nygaard I, DeLancey JO, Arnsdorf L, Murphy E. Exercise and incontinence. Obstet Gynecol. 1990 May;75(5):848-51. PMID 2325968
- [Background] Zhao B, Wen L, Liu D, Huang S. Urethral configuration and mobility during urine leaking described using real-time transperineal ultrasonography. Ultrasonography. 2022 Jan;41(1):171-176. doi: 10.14366/usg.21058. Epub 2021 Jun 15. PMID 34399041
- [Background] Zhang Y, Weaver RG, Armstrong B, Burkart S, Zhang S, Beets MW. Validity of Wrist-Worn photoplethysmography devices to measure heart rate: A systematic review and meta-analysis. J Sports Sci. 2020 Sep;38(17):2021-2034. doi: 10.1080/02640414.2020.1767348. Epub 2020 Jun 19. PMID 32552580
- [Background] Youssef A, Montaguti E, Sanlorenzo O, Cariello L, Salsi G, Morganelli G, Azzarone C, Pilu G, Rizzo N. Reliability of new three-dimensional ultrasound technique for pelvic hiatal area measurement. Ultrasound Obstet Gynecol. 2016 May;47(5):629-35. doi: 10.1002/uog.14933. Epub 2016 Mar 29. PMID 26105710
- [Background] Weinstein MM, Jung SA, Pretorius DH, Nager CW, den Boer DJ, Mittal RK. The reliability of puborectalis muscle measurements with 3-dimensional ultrasound imaging. Am J Obstet Gynecol. 2007 Jul;197(1):68.e1-6. doi: 10.1016/j.ajog.2007.02.041. PMID 17618762
- [Background] Teixeira RV, Colla C, Sbruzzi G, Mallmann A, Paiva LL. Prevalence of urinary incontinence in female athletes: a systematic review with meta-analysis. Int Urogynecol J. 2018 Dec;29(12):1717-1725. doi: 10.1007/s00192-018-3651-1. Epub 2018 Apr 13. PMID 29654349
- [Background] Serdar CC, Cihan M, Yucel D, Serdar MA. Sample size, power and effect size revisited: simplified and practical approaches in pre-clinical, clinical and laboratory studies. Biochem Med (Zagreb). 2021 Feb 15;31(1):010502. doi: 10.11613/BM.2021.010502. Epub 2020 Dec 15. PMID 33380887
- [Background] Schnider P, Birner P, Gendo A, Ratheiser K, Auff E. Bladder volume determination: portable 3-D versus stationary 2-D ultrasound device. Arch Phys Med Rehabil. 2000 Jan;81(1):18-21. doi: 10.1016/s0003-9993(00)90215-6. PMID 10638870
- [Background] Scherr J, Wolfarth B, Christle JW, Pressler A, Wagenpfeil S, Halle M. Associations between Borg's rating of perceived exertion and physiological measures of exercise intensity. Eur J Appl Physiol. 2013 Jan;113(1):147-55. doi: 10.1007/s00421-012-2421-x. Epub 2012 May 22. PMID 22615009
- [Background] Schallom M, Prentice D, Sona C, Vyers K, Arroyo C, Wessman B, Ablordeppey E. Accuracy of Measuring Bladder Volumes With Ultrasound and Bladder Scanning. Am J Crit Care. 2020 Nov 1;29(6):458-467. doi: 10.4037/ajcc2020741. PMID 33130866
- [Background] Pires T, Pires P, Moreira H, Viana R. Prevalence of Urinary Incontinence in High-Impact Sport Athletes: A Systematic Review and Meta-Analysis. J Hum Kinet. 2020 Jul 21;73:279-288. doi: 10.2478/hukin-2020-0008. eCollection 2020 Jul. PMID 32774559
- [Background] de Mattos Lourenco TR, Matsuoka PK, Baracat EC, Haddad JM. Urinary incontinence in female athletes: a systematic review. Int Urogynecol J. 2018 Dec;29(12):1757-1763. doi: 10.1007/s00192-018-3629-z. Epub 2018 Mar 19. PMID 29552736
- [Background] Hajebrahimi S, Nourizadeh D, Hamedani R, Pezeshki MZ. Validity and reliability of the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form and its correlation with urodynamic findings. Urol J. 2012 Fall;9(4):685-90. PMID 23235974
- [Background] Goldstick O, Constantini N. Urinary incontinence in physically active women and female athletes. Br J Sports Med. 2014 Feb;48(4):296-8. doi: 10.1136/bjsports-2012-091880. Epub 2013 May 18. PMID 23687004
- [Background] Gillinov S, Etiwy M, Wang R, Blackburn G, Phelan D, Gillinov AM, Houghtaling P, Javadikasgari H, Desai MY. Variable Accuracy of Wearable Heart Rate Monitors during Aerobic Exercise. Med Sci Sports Exerc. 2017 Aug;49(8):1697-1703. doi: 10.1249/MSS.0000000000001284. PMID 28709155
- [Background] Giagio S, Salvioli S, Innocenti T, Gava G, Vecchiato M, Pillastrini P, Turolla A. PFD-SENTINEL: Development of a screening tool for pelvic floor dysfunction in female athletes through an international Delphi consensus. Br J Sports Med. 2023 Jul;57(14):899-905. doi: 10.1136/bjsports-2022-105985. Epub 2022 Dec 14. PMID 36517214
- [Background] Giagio S. Bridging gaps, shaping futures: pelvic floor health for athletes (PhD Academy Award). Br J Sports Med. 2024 Jun 20;58(13):751-752. doi: 10.1136/bjsports-2024-108359. No abstract available. PMID 38724072
- [Background] Dietz HP, Rojas RG, Shek KL. Postprocessing of pelvic floor ultrasound data: how repeatable is it? Aust N Z J Obstet Gynaecol. 2014 Dec;54(6):553-7. doi: 10.1111/ajo.12250. Epub 2014 Oct 22. PMID 25338743
- [Background] Chan H. Noninvasive bladder volume measurement. J Neurosci Nurs. 1993 Oct;25(5):309-12. doi: 10.1097/01376517-199310000-00007. PMID 8270812
- [Background] Brown WJ, Miller YD. Too wet to exercise? Leaking urine as a barrier to physical activity in women. J Sci Med Sport. 2001 Dec;4(4):373-8. doi: 10.1016/s1440-2440(01)80046-3. PMID 11905931
- [Background] Bo K. Urinary incontinence, pelvic floor dysfunction, exercise and sport. Sports Med. 2004;34(7):451-64. doi: 10.2165/00007256-200434070-00004. PMID 15233598
- [Background] Yoshida S, Orimoto N, Tsukihara H, Noma T, Hakozaki A, Sasaki E. TAC-302 promotes neurite outgrowth of isolated peripheral neurons and prevents bladder denervation related bladder dysfunctions following bladder outlet obstruction in rats. Neurourol Urodyn. 2018 Feb;37(2):681-689. doi: 10.1002/nau.23375. Epub 2017 Jul 26. PMID 28745805